CLINICAL TRIAL: NCT04433221
Title: Safety and Efficacy Evaluation of a Combination Immunotherapy Targeting Sarcomas
Brief Title: Combination Immunotherapy Targeting Sarcomas
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Collaborators: The Seventh Affiliated Hospital of Sun Yat-sen University (Other); Shenzhen Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-20007
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Sarcoma; Osteoid Sarcoma; Ewing Sarcoma
Keywords: Sarcoma; Chemotherapy; Doxorubicin; CART; Vaccine
MeSH Terms: conditions — Sarcoma; Bone Neoplasms; Sarcoma, Ewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multiple sarcoma-specific CAR-T cells (Experimental): Patients who have confirmed surface antigens including GD2, PSMA, Her2, CD276 or other markers
  Interventions: Biological: Multiple sarcoma-specific CAR-T cells and sarcoma vaccines

INTERVENTIONS:
Biological: Multiple sarcoma-specific CAR-T cells and sarcoma vaccines — 1 infusion, CART 1x10^6~1x10^7 cells/kg via IV and vaccines 1-5x10^6 irradiated cells via subcutaneous injection

SUMMARY:
The aim of this clinical trial is to assess the feasibility, safety and efficacy of a combination low dose chemotherapy and immunotherapy in patients who have sarcoma that is relapsed or late staged. Another goal of the study is to assess the safety and efficacy of the therapy that combines multiple CAR T cells followed by sarcoma vaccines.

DETAILED DESCRIPTION:
Patients with late staged and/or recurrent sarcoma have poor prognosis despite complex multimodal therapy. Therefore, innovative interventions are needed. Sarcoma is known to express increased levels of surface antigens that can be targeted by CAR-T cells. In addition, studies have shown that low dose chemotherapy such as doxorubicin may modulate surface PD-L1 level and enhance immunotherapy effects. This study will combine multiple CAR T cells with low dose chemotherapy to treat sarcoma, and followed by maintenance sarcoma vaccines. The purpose of this clinical trial will assess the feasibility, safety, efficacy and side effects of this combination therapy in patients who have sarcoma that is relapsed or late staged.

ELIGIBILITY:
Inclusion Criteria:

1. Stage Ⅲ，Ⅳ sarcoma patients or recurrent sarcoma patients;
2. Age: ≥ 6 months and ≤80 years of age at the time of enrollment;
3. At least 2 weeks since the last standard chemotherapy or radiotherapy and immunosuppressive therapy such as steroid hormone before enrollment;
4. Side effects of chemotherapy have been well managed;
5. Confirmed malignant cell expression of CART target antigens by IHC or flow
6. Karnofsky /jansky score of 50% or greater;
7. Expected survival > 8 weeks;
8. ANC≥ 1×10^6/L，PLT ≥ 1×10^8/L;
9. Pulse oximetry of≥90% on room air；
10. Adequate hepatic function, defined as aspartate aminotransferase(AST)< 5 times upper limit of normal(ULN),serum bilirubin < 3 times ULN;
11. Adequate renal function, defined as serum creatinine less than 2 times ULN, if serum creatinine more than 1.5 times ULN, creatinine clearance rate test is needed;
12. Patients must have sufficient autologous CART cells at does greater than 0.5x10^6 cells/kg body weight;
13. Sign an informed consent and assent.

Exclusion Criteria:

1. The disease is progressing rapidly;
2. The patient is receiving therapy of other new drugs and under evaluation;
3. Evidence of tumor potentially causing airway obstruction;
4. Epilepsy history or other CNS diseases;
5. Patients who need immunosuppressive drugs;
6. History of long QT syndrome or severe heart diseases;
7. Uncontrolled active infection;
8. Active hepatitis B virus, hepatitis C virus or HIV infection;
9. Receiving systemic corticosteroid 2 weeks before enrollment except for inhaled steroids;
10. Previous treatment with any gene therapy;
11. Creatinine>2.5mg/dl or ALT/AST>3 times normal or bilirubin>2.0 mg/dl;
12. Patients who have other uncontrolled diseases such as obstruction of lung function would preclude participation as outlined;
13. Pregnant or lactating women;
14. Patients previously experienced toxicity from cyclophosphamide and doxorubicin;
15. Patients who have CNS sarcoma;
16. In condition that may bring risks to subjects or interference to clinical trials.

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of CART cells infusion | 3 months
  Safety of CART cells in patients using CTCAE version 4.0 standard to evaluate the level of adverse events

SECONDARY OUTCOMES:
Overall survival Rate | 1 year
  Percentage of participants with objective response as determined by the investigator based on Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1)
Treatment response rate of sarcomas | 1 year
  Defined as the proportion of patients who achieved complete remission (CR), partial remission (PR), stable disease (SD), or progressive disease (PD) based on CT imaging analysis.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shenzhen Children's Hospital, Shenzhen, Guangdong
  - The Seventh Affilliated Hospital, Sun Yat-Sen University, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: No